CLINICAL TRIAL: NCT03073980
Title: Assessing Efficacy of Intravenous Acetaminophen for Perioperative Pain Control for Oocyte Retrieval: a Randomized, Double Blind, Placebo-controlled Trial
Brief Title: Assessing Efficacy of Intravenous Acetaminophen for Perioperative Pain Control for Oocyte Retrieval
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, John C Petrozza, Chief, Division of Reproductive Medicine and IVF, Principal Investigator, Clinical Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016P002465
Record Dates: First submitted 2017-02-22; First posted 2017-03-08 (Actual); Results first posted 2022-04-20 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Infertility, Female; Pain, Postoperative
Keywords: in vitro fertilization; oocyte retrieval; acetaminophen; postoperative pain control
MeSH Terms: conditions — Infertility, Female; Pain, Postoperative | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Intravenous (IV) acetaminophen/oral (PO) placebo (Experimental): In the pre-operative suite, these patients will receive 1000mg IV acetaminophen and PO placebo, followed by standard protocol anesthesia and pain control as needed.
  Interventions: Drug: IV Acetaminophen; Other: Placebo PO Acetaminophen
- Group 2: Intravenous (IV) placebo/oral (PO) acetaminophen (Active Comparator): In the pre-op suite, these patients will receive 1000mg PO acetaminophen and IV placebo, followed by standard protocol anesthesia and pain control as needed.
  Interventions: Drug: PO Acetaminophen; Other: Placebo IV Acetaminophen
- Group 3: Oral and intravenous Placebo / Standard of care (Placebo Comparator): In the pre-op suite, these patients will receive PO and IV placebo, followed by standard protocol anesthesia and pain control as needed.
  Interventions: Other: Placebo IV Acetaminophen; Other: Placebo PO Acetaminophen

INTERVENTIONS:
Drug: IV Acetaminophen — IV Acetaminophen for pain control during procedure
  Arms: Group 1: Intravenous (IV) acetaminophen/oral (PO) placebo
Drug: PO Acetaminophen — PO Acetaminophen for pain control during procedure
  Arms: Group 2: Intravenous (IV) placebo/oral (PO) acetaminophen
Other: Placebo IV Acetaminophen — Placebo IV Acetaminophen
  Arms: Group 2: Intravenous (IV) placebo/oral (PO) acetaminophen; Group 3: Oral and intravenous Placebo / Standard of care
Other: Placebo PO Acetaminophen — Placebo PO Acetaminophen
  Arms: Group 1: Intravenous (IV) acetaminophen/oral (PO) placebo; Group 3: Oral and intravenous Placebo / Standard of care

SUMMARY:
In this research study we want to learn more about how effective certain medications are at reducing pain after oocyte (egg) retrieval surgery and how effective they are at reducing the time between the retrieval and discharge from the hospital. We will compare three types of pre-operative medications: intravenous (IV) acetaminophen, oral (PO) acetaminophen, and placebo (no medication), which is the current typical care.

DETAILED DESCRIPTION:
OBJECTIVE: To compare the efficacy of pre-operative IV acetaminophen, PO acetaminophen, versus placebo for adjunctive pain control in the setting of oocyte retrieval in an in vitro fertilization clinic setting.

HYPOTHESIS: Our hypothesis is that patients receiving IV acetaminophen pre-operatively will have improved postoperative pain scores, lower overall opiate consumption, and shortened time to discharge from post analgesic recovery unit (PACU) or recovery than those receiving PO acetaminophen or placebo.

Participants will be consented and enrolled in the study prior to their oocyte retrieval. The patient will then be randomized to one of three treatments:

Group 1: In the pre-op suite, these patients will receive 1000mg IV acetaminophen and PO placebo, followed by standard protocol anesthesia and pain control as needed.

Group 2: In the pre-op suite, these patients will receive 1000mg PO acetaminophen and IV placebo, followed by standard protocol anesthesia and pain control as needed.

Group 3:

In the pre-op suite, these patients will receive PO and IV placebo, followed by standard protocol anesthesia and pain control as needed.

The patient and care team will be blinded to the treatment group.

A member of the study staff will review participants' medical record to collect data regarding demographics, clinical history, cycle and pregnancy outcomes, up to 12 months following study completion.

ELIGIBILITY:
Inclusion Criteria:

[ ] Patient is 18 years or over, undergoing oocyte retrieval. [ ] Patient is English-speaking.

Exclusion Criteria:

[ ] Allergy/hypersensitivity to acetaminophen or opiates. [ ] Any history of liver disease, history of alcohol depending, or renal impairment as reported in the electronic health record.

[ ] Any history chronic opiate use or chronic pain disorder reported in the electronic health record.

[ ] Weight less than 50kg as reported in the medical record.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Petrozza, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sacha CR, Mortimer R, Hariton E, James K, Hosseini A, Gray M, Xuan C, Hammer K, Lange A, Mahalingaiah S, Wang J, Petrozza JC. Assessing efficacy of intravenous acetaminophen for perioperative pain control for oocyte retrieval: a randomized, double-blind, placebo-controlled trial. Fertil Steril. 2022 Jan;117(1):133-141. doi: 10.1016/j.fertnstert.2021.08.046. Epub 2021 Sep 20. PMID 34548165

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: IV Acetaminophen/PO Placebo: In the pre-op suite, these patients will receive 1000mg IV acetaminophen and PO placebo, followed by standard protocol anesthesia and pain control as needed.
  IV Acetaminophen: IV Acetaminophen for pain control during procedure
  Placebo PO Acetaminophen: Placebo PO Acetaminophen
- Group B: IV Placebo/PO Acetaminophen: In the pre-op suite, these patients will receive 1000mg PO acetaminophen and IV placebo, followed by standard protocol anesthesia and pain control as needed.
  PO Acetaminophen: PO Acetaminophen for pain control during procedure
  Placebo IV Acetaminophen: Placebo IV Acetaminophen
- Group C: IV Placebo/ PO Placebo: In the pre-op suite, these patients will receive PO and IV placebo, followed by standard protocol anesthesia and pain control as needed.
  Placebo IV Acetaminophen: Placebo IV Acetaminophen
  Placebo PO Acetaminophen: Placebo PO Acetaminophen
Period: Overall Study
Arm/Group | Group A: IV Acetaminophen/PO Placebo | Group B: IV Placebo/PO Acetaminophen | Group C: IV Placebo/ PO Placebo
Started | 53 | 54 | 54
Completed | 43 | 52 | 43
Not Completed | 10 | 2 | 11
Not completed — Lost to Follow-up | 10 | 2 | 9
Not completed — No post-procedure data | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Group C: IV Placebo / PO Placebo: In the pre-op suite, these patients will receive PO and IV placebo, followed by standard protocol anesthesia and pain control as needed.
  Placebo IV Acetaminophen: Placebo IV Acetaminophen
  Placebo PO Acetaminophen: Placebo PO Acetaminophen
- Total: Total of all reporting groups
Arm/Group | Group A: IV Acetaminophen/PO Placebo | Group B: IV Placebo/PO Acetaminophen | Group C: IV Placebo / PO Placebo | Total
Number analyzed (Participants) | 53 | 54 | 52 | 159
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 53 | 54 | 52 | 159
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (4.1) | 35.7 (4.5) | 36.0 (4.0) | 35.6 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 54 | 52 | 159
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4 | 8
  Not Hispanic or Latino | 2 | 3 | 2 | 7
  Unknown or Not Reported | 48 | 50 | 46 | 144
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 4 | 6 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 5
  White | 41 | 43 | 39 | 123
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 5 | 6 | 16
Region of Enrollment [Number; unit: participants]
  United States | 53 | 54 | 52 | 159
Ovarian reserve (anti-mullerian hormone) [Mean (Standard Deviation); unit: ng/ml] | 2.9 (2.9) | 3.0 (2.4) | 2.4 (1.7) | 2.8 (2.3)
Number of Nulliparous Participants [Number; unit: Participants] | 41 | 39 | 43 | 123
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.4 (4.7) | 24.9 (4.1) | 25.6 (4.9) | 25.3 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain Score Difference 10 Mins From Pre-operative
Description: Visual analog scale of pain, ranging from 0 (no pain) to 10 (worst pain imaginable) in whole numbers. The final score is the post-operative score minus the pre-operative score.
Time Frame: Pain was measured pre-operatively and at 10 minutes post-procedure.
Population: Post-operative pain score - pre-operative pain score; 2 patients in group 3 had egg retrieval cancelled due to Coronavirus Disease (COVID); data could not be collected in these patients, yet their enrollment was included in an intention-to-treat analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Group 1: IV Acetaminophen/PO Placebo: In the pre-op suite, these patients will receive 1000mg IV acetaminophen and PO placebo, followed by standard protocol anesthesia and pain control as needed.
  IV Acetaminophen: IV Acetaminophen for pain control during procedure
  Placebo PO Acetaminophen: Placebo PO Acetaminophen
- Group 2: IV Placebo/PO Acetaminophen: In the pre-op suite, these patients will receive 1000mg PO acetaminophen and IV placebo, followed by standard protocol anesthesia and pain control as needed.
  PO Acetaminophen: PO Acetaminophen for pain control during procedure
  Placebo IV Acetaminophen: Placebo IV Acetaminophen
- Group 3: IV Placebo/PO Placebo: In the pre-op suite, these patients will receive PO and IV placebo, followed by standard protocol anesthesia and pain control as needed.
  Placebo IV Acetaminophen: Placebo IV Acetaminophen
  Placebo PO Acetaminophen: Placebo PO Acetaminophen
Arm/Group | Group 1: IV Acetaminophen/PO Placebo | Group 2: IV Placebo/PO Acetaminophen | Group 3: IV Placebo/PO Placebo
Number analyzed (Participants) | 53 | 54 | 52
score on a scale | 1.3 (2.4) | 1.3 (2.8) | 1.8 (1.8)

2. Primary Outcome: Time to Discharge From the Post-operative Recovery Room
Description: Discharge time was based on the nurse's assessment of patient alertness, ability to tolerate oral liquids and food, and ability to void.
Time Frame: 0-6 hours post-procedure
Population: 2 patients in group 3 had egg retrieval cancelled due to COVID; data could not be collected in these patients, yet their enrollment was included in an intention-to-treat analysis.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Group 3: Placebo / Standard of Care: In the pre-op suite, these patients will receive PO and IV placebo, followed by standard protocol anesthesia and pain control as needed.
  Placebo IV Acetaminophen: Placebo IV Acetaminophen
  Placebo PO Acetaminophen: Placebo PO Acetaminophen
Arm/Group | Group 1: IV Acetaminophen/PO Placebo | Group 2: IV Placebo/PO Acetaminophen | Group 3: Placebo / Standard of Care
Number analyzed (Participants) | 53 | 54 | 52
minutes | 60.1 (22.0) | 58.8 (17.0) | 57.6 (10.7)

3. Secondary Outcome: Procedure Length
Description: Duration of egg retrieval
Time Frame: 0-2 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group A: IV Acetaminophen/PO Placebo | Group B: IV Placebo/PO Acetaminophen | Group C: IV Placebo/ PO Placebo
Number analyzed (Participants) | 53 | 54 | 52
minutes | 13.5 (5.9) | 13.7 (5.3) | 14.1 (6.6)

4. Secondary Outcome: Postoperative Nausea and Vomiting
Description: One or more episodes of nausea and vomiting in the recovery room and through post-operative day 2
Time Frame: 0-2 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: IV Acetaminophen/PO Placebo | Group B: IV Placebo/PO Acetaminophen | Group C: IV Placebo/ PO Placebo
Number analyzed (Participants) | 53 | 54 | 52
Participants | 3 | 4 | 2

5. Secondary Outcome: Oocyte Yield
Description: The number of oocytes retrieved from the patient's ovaries as part of an in vitro-fertilization treatment. This includes both immature and mature oocytes.
Time Frame: 0 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | Group A: IV Acetaminophen/PO Placebo | Group B: IV Placebo/PO Acetaminophen | Group C: IV Placebo/ PO Placebo
Number analyzed (Participants) | 53 | 54 | 52
oocytes | 12.6 (8.8) | 13.4 (8.7) | 11.4 (5.9)

6. Secondary Outcome: Rescue Medication Required
Description: One or more doses of opiate pain medication given due to pain during the procedure or immediately post-operative in the recovery room.
Time Frame: During procedure and immediately post-operative in recovery room within 45 minutes
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: IV Acetaminophen/PO Placebo | Group B: IV Placebo/PO Acetaminophen | Group C: IV Placebo/ PO Placebo
Number analyzed (Participants) | 53 | 54 | 52
Participants | 4 | 10 | 8

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Data was collected during procedural period, post-procedure, and during embryo development and 1st 12 weeks of pregnancy
Arm/Group | Group A: IV Acetaminophen/PO Placebo | Group B: IV Placebo/PO Acetaminophen | Group C: IV Placebo/ PO Placebo
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/54 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 0/53 | 0/54 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT03073980/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/80/NCT03073980/ICF_001.pdf